CLINICAL TRIAL: NCT05557396
Title: The Efficiency of Internal Tube Length Measurement Methods in Correct Placement of the Nasogastric Tube
Brief Title: Internal Tube Length of the Nasogastric Tube
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The targeted sample size could not be reached
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nihal Taskiran, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: nasogastric tube
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Feeding Tube Complication
Keywords: nasogastric tube; internal tube length; critical care; nursing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- NEX (Control group) (Active Comparator): Nose-ear-xiphoid measurement method (NEX), (n=31)
  The distance between the patient's nose tip and earlobe will be measured first, then the distance between the earlobe and the xiphoid (NEX method) Marking will be made on the nasogastric tube according to the length obtained from the measurement, The nasogastric tube will be advanced by the researcher from the patient's nose to the point where the marking is made, Immediately after the completion of the nasogastric tube placement procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
  Interventions: Other: Internal Tube Length Measurement Procedures for Nazogastric Tube
- CoNEX (Experimental): Corrected nose-earlobe-xiphoid measurement method (CoNEX), (n=31) The distance between the patient's nose tip and earlobe will be measured first, and then the distance between the earlobe and the xiphoid, The nasogastric tube length to be applied to the patient will be determined according to the formula (NEX x 0.38696) + 36.37 cm, The length determined according to the result obtained will be marked on the nasogastric tube, The nasogastric tube will be advanced by the researcher from the patient's nose to the point where the marking is made, Immediately after the completion of the nasogastric tube placement procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
  Interventions: Other: Internal Tube Length Measurement Procedures for Nazogastric Tube
- XEN+10 (Experimental): Xiphoid-earlobe-nose+10 cm (XEN+10), (n=31)
  The distance between the patient's xiphoid and earlobe will be measured first, and then the distance between the earlobe and the tip of the nose will be measured and 10 cm will be added to the obtained measurement, The length determined according to the result obtained will be marked on the nasogastric tube, The nasogastric tube will be advanced by the researcher from the patient's nose to the point where the marking is made, Immediately after the completion of the nasogastric tube placement procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
  Interventions: Other: Internal Tube Length Measurement Procedures for Nazogastric Tube
- GWNUF (Experimental): Gender-weight-nose-umblikus-head flat (GWNUF), (n=31)
  The patient's body weight will be measured without clothes on, When the patient is in the supine position, the distance between the tip of the nose and the umbilicus will be measured, The length of the nasogastric tube to be applied to the patient according to the formula 29.38 + (4.53 x gender) + (0.34 x distance between the tip of the nose and the umbilicus) - (0.06 x patient weight), (gender = 1 for male patient, 0 for female patient) to be determined, The length determined according to the result obtained will be marked on the nasogastric tube, The nasogastric tube will be advanced by the researcher from the patient's nose to the point where the marking is made, Immediately after the completion of the insertion procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
  Interventions: Other: Internal Tube Length Measurement Procedures for Nazogastric Tube
- EXU-NE (Experimental): The distance between the patient's xiphoid and earlobe will be measured first (Measurement 1), (n=31) The distance between the patient's xiphoid and the midline of the umbilicus will be measured (Measurement 2), The two obtained measurement values will be added (Measurement 1 + Measurement 2), The distance between the patient's nose tip and earlobe will be measured (Measurement 3), Measurement 3 value will be subtracted from the sum of Measurement 1 and Measurement 2 values, The length determined according to the result obtained will be marked on the nasogastric tube, The nasogastric tube will be advanced by the researcher from the patient's nose to the point where the marking is made, Immediately after the completion of the insertion procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
  Interventions: Other: Internal Tube Length Measurement Procedures for Nazogastric Tube

INTERVENTIONS:
Other: Internal Tube Length Measurement Procedures for Nazogastric Tube — Different Internal Tube Length Measurement Procedures will used for the correct placement of nasogastric tube.

SUMMARY:
This methodological research is aimed to examine the effectiveness of the methods used to estimate the internal length of the nasogastric tube and to determine the most reliable method for correct placement of the nasogastric tube in adults.

The study will be carried out between 01 September 2022 and 01 September 2023 with 155 patients who hospitalized in the anesthesia and reamination intensive care and general intensive care units of Aydın Adnan Menderes University Application and Research Hospital.

The internal tube length measurement methodologies will utilized to confirm proper NGT placement. A total of 5 groups will be included in the study, including 1 control (NEX measurement method) and 4 experimental groups, (Experiment 1: CoNEX measurement method, Experiment 2: XEN+10 cm measurement method, Experiment 3: GWNUF measurement method, Experiment 4: EXU-NE Method measurement method).The "gold standard" reference method will used for comparison was radiography.

Research data will be analyzed in SPSS (Statistical Package for Social Sciences) for Windows 25.0 statistical package program. Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of the data. The comparison between the methods used in the measurement of the nasogastric tube (NEX, CoNEX, XEN+10 cm, GWNUF, EXU-NE) and the results of the radiological evaluation (reference method) will be made with Chi-square analysis. Statistical significance will be accepted as p<0.05.

DETAILED DESCRIPTION:
This research is a methodological study in a single-blind randomized controlled experimental model. This research is aimed to examine the effectiveness of the methods used to estimate the internal length of the nasogastric tube and to determine the most reliable method for correct placement of the nasogastric tube in adults.

The study will be carried out between September 2022-September 2023 with 155 patients who hospitalized in the anesthesia and reamination intensive care and general intensive care units of Aydın Adnan Menderes University Application and Research Hospital.

A total of five internal tube length measurement methodologies will utilized to determine the length of NGT to be placed on the patient. These methods are CoNEX measurement method (Experiment 1), XEN+10 cm measurement method (Experiment 2), GWNUF measurement method (Experiment 3), EXU-NE Method measurement method (Experiment 4) and NEX measurement method (control). To collect data, a ''Case Report Form'' is carried out. This form consisted of 17 items regarding each patient's descriptive characteristics (age, gender, etc.), data concerning their illness and treatment (duration in intensive care, medical diagnosis, existing chronic disease, level of consciousness, drugs being administered) as well as data about the NGT intubation (type and gauge of NGT, observation for signs of respiratory distress, other complications, etc.).Patient information will obtained from their medical records. All the NGT placements will conducted by the same researcher under the supervision of the other two researchers. Following NGT insertion, "abdominal x-ray"(gold standard)" reference method will used to confirm the placement of NGT.

Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of the data. The comparison between the methods used in the measurement of the nasogastric tube (NEX, CoNEX, XEN+10 cm, GWNUF, EXU-NE) and the results of the radiological evaluation (reference method) will be made with Chi-square analysis. Statistical significance will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* >18 age,
* Being a patient in the adult intensive care units of the hospital where the research was conducted,
* Glasgow coma scale ≤8,

Exclusion Criteria:

* Patients fed through orogastric, orojejunal, gastrostomy, jegenostomy, and ostomy,
* Patients who are pregnant or suspected of pregnancy,
* Patients presenting with a history of trauma,
* Patients with esophageal varices, nasal septal deviation, upper respiratory tract and/or digestive system anomalies,
* Patients who had a nasogastric tube inserted or whose nasogastric tube would be changed before participating in the study,
* Patients whose nose-earlobe-xiphoid distance cannot be measured,
* Patients who are not accepted to participate in the study by their legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The CoNEX method is an effective measurement method to accurately determine the internal length of the nasogastric tube. | One year
  By creating a straight line with a tape measure, first the distance between the patient's nose tip and the earlobe and then the distance between the earlobe and the xiphoid will be measured, then the nasogastric tube length to be applied to the patient will be determined according to the (NEX x 0.38696) + 36.37 cm formula. The length determined according to the result will be marked on the nasogastric tube, and the nasogastric tube will be advanced by the researcher from the patient's nose to the marked place.Immediately after the completion of the insertion process, an abdominal X-ray will be taken and the tube location will be confirmed.
The XEN+10 cm method is an effective measurement method to accurately determine the internal length of the nasogastric tube. | one year
  By creating a straight line with a tape measure, the distance between the patient's xiphoid and earlobe, then the distance between the earlobe and the tip of the nose will be measured and 10 cm will be added to the measurement obtained. The location of the tube will be confirmed by taking an abdominal x-ray immediately after the placement process is completed, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
The GWNUF method is an effective measurement method to accurately determine the internal length of the nasogastric tube. | one year
  Body weight will be measured without clothing on the patient, The distance between the tip of the nose and the umbilicus will be measured while the patient is in the supine position, 29.38 + (4.53 x gender) + (0.34 x distance between the tip of the nose and the umbilicus) - (0.06 x patient weight), (gender) The length of the nasogastric tube to be applied to the patient will be determined according to the formula = 1 for male patient, 0 for female patient, The length determined according to the result obtained will be marked on the nasogastric tube, The nasogastric tube will be advanced by the investigator from the patient's nose to the marked area, Immediately after the completion of the insertion procedure, the abdominal X-ray will be determined. The tube location will be confirmed by filming, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
EXU-NE method is an effective measurement method to accurately determine the internal length of the nasogastric tube. | One year
  By creating a straight line with a tape measure, the distance between the patient's xiphoid and earlobe will be measured first (Measurement 1), The distance between the patient's xiphoid and the midline of the umbilicus will be measured (Measure 2), The two obtained measurement values will be added (Measurement 1 + Measurement 2), The distance between the patient's nose tip and earlobe will be measured (Measurement 3), Measurement 3 value will be subtracted from the sum of Measurement 1 and Measurement 2 values, The length determined according to the result obtained will be marked on the nasogastric tube, The nasogastric tube will be advanced by the researcher from the patient's nose to the marked place, Insertion Immediately after the completion of the procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.
The NEX method is an effective measurement method to accurately determine the internal length of the nasogastric tube. | One year
  By creating a straight line with a tape measure, first the distance between the patient's nose tip and the earlobe and then the distance between the earlobe and the xiphoid will be measured, A marking will be made on the nasogastric tube according to the length obtained from the measurement, The nasogastric tube will be advanced by the researcher from the patient's nose to the point where the marking is made, Immediately after the completion of the nasogastric tube placement procedure, an abdominal X-ray will be taken to confirm the tube location, the position of the distal end of the tube relative to the gastro-esophageal junction will be measured and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Taskiran, PhD, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Nihal Taskiran-study protocol Pakize Özçiftçi Yılmaz-informed consest form Dilek Sarı-Statistical analysis plan Tuna Şahin_study protocol Necla Olcum- informed consent form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one year
Access Criteria: Reaching the target sample size

REFERENCES:
- [Result] Chen YC, Wang LY, Chang YJ, Yang CP, Wu TJ, Lin FR, Liu SY, Wei TS. Potential risk of malposition of nasogastric tube using nose-ear-xiphoid measurement. PLoS One. 2014 Feb 10;9(2):e88046. doi: 10.1371/journal.pone.0088046. eCollection 2014. PMID 24520344
- [Result] Best C. How to insert a nasogastric tube and check gastric position at the bedside. Nurs Stand. 2016 May 18;30(38):36-40. doi: 10.7748/ns.30.38.36.s43. PMID 27191450
- [Result] Santos SC, Woith W, Freitas MI, Zeferino EB. Methods to determine the internal length of nasogastric feeding tubes: An integrative review. Int J Nurs Stud. 2016 Sep;61:95-103. doi: 10.1016/j.ijnurstu.2016.06.004. Epub 2016 Jun 15. PMID 27328376
- [Result] Ellett ML, Cohen MD, Perkins SM, Croffie JM, Lane KA, Austin JK. Comparing methods of determining insertion length for placing gastric tubes in children 1 month to 17 years of age. J Spec Pediatr Nurs. 2012 Jan;17(1):19-32. doi: 10.1111/j.1744-6155.2011.00302.x. Epub 2011 Sep 30. PMID 22188269
- [Result] Ellett ML, Beckstrand J, Flueckiger J, Perkins SM, Johnson CS. Predicting the insertion distance for placing gastric tubes. Clin Nurs Res. 2005 Feb;14(1):11-27; discussion 28-31. doi: 10.1177/1054773804270919. PMID 15604226
- [Result] Fan PEM, Tan SB, Farah GI, Cheok PG, Chock WT, Sutha W, Xu D, Chua W, Kwan XL, Li CL, Teo WQ, Ang SY. Adequacy of different measurement methods in determining nasogastric tube insertion lengths: An observational study. Int J Nurs Stud. 2019 Apr;92:73-78. doi: 10.1016/j.ijnurstu.2019.01.003. Epub 2019 Jan 14. PMID 30743198
- [Result] Malta MA, Carvalho-Junior AF, Andreollo NA, Freitas MI. [Anthropometric measures for the introduction of the nasogastric tube for enteral nutrition employing the esophagogastroduodenoscopy]. Arq Bras Cir Dig. 2013 Jun;26(2):107-11. doi: 10.1590/s0102-67202013000200007. Portuguese. PMID 24000021
- [Result] Taylor SJ, Allan K, McWilliam H, Toher D. Nasogastric tube depth: the 'NEX' guideline is incorrect. Br J Nurs. 2014 Jun 26-Jul 9;23(12):641-4. doi: 10.12968/bjon.2014.23.12.641. PMID 25039627
- [Result] Taylor SJ. Methods of Estimating Nasogastric Tube Length: All, Including "NEX," Are Unsafe. Nutr Clin Pract. 2020 Oct;35(5):864-870. doi: 10.1002/ncp.10497. Epub 2020 May 14. PMID 32406552
- [Result] Torsy T, Saman R, Boeykens K, Duysburgh I, Eriksson M, Verhaeghe S, Beeckman D. Accuracy of the corrected nose-earlobe-xiphoid distance formula for determining nasogastric feeding tube insertion length in intensive care unit patients: A prospective observational study. Int J Nurs Stud. 2020 Oct;110:103614. doi: 10.1016/j.ijnurstu.2020.103614. Epub 2020 May 11. PMID 32702567
- [Result] Torsy T, Saman R, Boeykens K, Duysburgh I, Van Damme N, Beeckman D. Comparison of Two Methods for Estimating the Tip Position of a Nasogastric Feeding Tube: A Randomized Controlled Trial. Nutr Clin Pract. 2018 Dec;33(6):843-850. doi: 10.1002/ncp.10112. Epub 2018 Jun 30. PMID 29959848